CLINICAL TRIAL: NCT03596190
Title: Diaphragmatic Dysfunction After Ultrasound-guided Supraclavicular Brachial Plexus Block With the Double Injection Technique
Brief Title: Diaphragmatic Dysfunction After Supraclavicular Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Vishal Uppal, Principal Investigator, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6447
Record Dates: First submitted 2018-06-04; First posted 2018-07-23 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessment arm (Other)
  Interventions: Diagnostic Test: ultrasonographic diaphragmatic assessment

INTERVENTIONS:
Diagnostic Test: ultrasonographic diaphragmatic assessment — Diaphragmatic dysfunction will be determined by intercostal diaphragm thickening. The available image will be saved.
  Diaphragmatic motion assessments will be conducted on the side to be blocked both at baseline, and then every 5 minutes until patient leaves for operating room or 30 minutes (whatever is earlier).

SUMMARY:
The investigators plan to determine the onset time and incidence of hemidiaphragmatic paresis (HDP) with a double injection supraclavicular nerve block in patients presenting for upper extremity surgery below the elbow.

The hypothesis is HDP following supraclavicular brachial plexus block occurs with-in 15 minutes of block performance and is not associated with subjective dyspnea.

DETAILED DESCRIPTION:
This study will be an observational trial to assess the onset time and incidence of hemidiaphragmatic paresis in patients who undergo the double injection ultrasound-guided supraclavicular block. Diaphragmatic dysfunction will be determined by intercostal diaphragm thickening measured using ultrasound. The available image will be saved.

Patients having below the elbow surgery will be be approached by someone from the research team for consent and possible inclusion in the study. This will be done in the anesthesia preoperative assessment clinic, or in the pre-op area on the day of surgery (if a patient was not seen in clinic).

A baseline ultrasonographic diaphragmatic assessment will be completed. Study participants will then receive supraclavicular brachial plexus block as per standard of care. Ultrasonographic diaphragmatic assessment and dyspnea score (using modified Borg dyspnea scale) will be performed every 5 minutes for 30 minutes, or until the patient is transferred to the operating room, whatever comes first. Patients will also undergo an ultrasonographic diaphragmatic assessment and dyspnea score in the recovery room after their surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for unilateral upper extremity surgery below the level of the elbow (the forearm or hand) who are having a double injection regional block for anesthesia
* 18 years old and over
* Weight 50kg or greater
* English speaking
* American Society of Anesthesiologists physical status 1-3

Exclusion Criteria:

* Known Chronic Obstructive Pulmonary Disease
* Pregnancy
* Any significant neurologic dysfunction, or inability to visualize the diaphragm during baseline sonographic assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Frequency of hemi-diaphragmatic paresis | Relative change in ultrasound assessment of diaphragmatic thickening (Baseline vs 30 min after supraclavicular block)
  Number of participants in which hemi-diaphragmatic paresis is detected using ultrasound measurement of diaphragmatic thickening
Onset time of hemi-diaphragmatic paresis | Baseline, 5, 10, 15, 20, 25, and 30 minutes after block
  The average time at which hemi-diaphragmatic paresis is detected using ultrasound measurement of diaphragmatic thickening

SECONDARY OUTCOMES:
The correlation of subjective dyspnea | Baseline, 5, 10, 15, 20, 25, and 30 minutes after block
  Using the modified Borg dyspnea scale ranging from 0 (no breathlessness at all to 10 (maximal breathlessness)
Incidence of HDP after surgical procedure under supraclavicular brachial plexus block (in post recovery unit). | Post-operatively up to 24 hours
  Based upon sonographic assessment

CONTACTS AND LOCATIONS:
Locations (1):
- NSHA, Halifax, Nova Scotia, Canada